| DOCUMENT DATE (IRB APPROVAL): |
|---|
| 03-Jan-2024 |
| NCT NUMBER: |
| NCT05938816 |
| OFFICIAL STUDY TITLE: |
| Feasibility and acceptability of stress induction, physiological data collection, and Mindfulness-Based Stress Reduction among combat veterans with PTSD |
| INVESTIGATOR NAME: |
| Josh Kaplan, PhD, MCR |
| ORGANIZATION: |
| Oregon Health & Science University |

# 1) Protocol Title

Feasibility and acceptability of stress induction, physiological data collection, and Mindfulness-Based Stress Reduction among combat veterans with PTSD

# 2) Objectives

Objectives are to gather feasibility and acceptability of key study elements (e.g., stress induction via cognitive stressor, physiological data collection including respiration, blood pressure, and heart rate, and the target intervention Mindfulness-Based Stress Reduction) among combat veterans experiencing PTSD symptoms to support a future K23 grant resubmission. Specific Aims are as follows:

Aim 1: Assess feasibility and participant acceptability of intervention and randomization procedures. Aim 1A: Examine acceptability of MBSR via qualitative data gathered during a post-intervention focus group.

Aim 1B: Assess feasibility of recruiting and acceptability of randomizing participants to an MBSR or active control condition. Recruitment, differential retention, and home practice completion rates will be examined.

Aim 2: Assess feasibility and participant acceptability of concurrent stress induction and physiological data collection (i.e., systolic [SBP] and diastolic [DBP] blood pressure) procedures.

Aim 2A: Evaluate feasibility of stress induction via significant change in BP from baseline to stressor. Aim 2B: Examine acceptability of physiological data collection concurrent with stressor task via focus group.

Aim 3: Evaluate sensitivity and responsiveness to change of outcome measures. Examining these qualities and pre-post changes in physiological and psychological resilience and PTSD symptoms will provide crucial information regarding relationships between the intervention and changes in relevant variables.

# 3) Background

Posttraumatic stress disorder (PTSD) is a significant public health concern<sup>1</sup> that negatively impacts quality of life and functioning,<sup>1-3</sup> is associated with increased mortality,<sup>4</sup> and poses an economic burden.<sup>5</sup>

Practice Guidelines<sup>9</sup> recommend cognitive processing therapy (CPT) and prolonged exposure (PE). Although research supports these treatments, <sup>10-12</sup> they present significant shortcomings: (1) they may not be acceptable for all patients, <sup>13</sup> (2) they show attrition as high as 40%, <sup>14-16</sup> and (3) they often result in residual symptoms. <sup>7,8</sup> Symptoms such as higher physiological arousal <sup>17,18</sup> and stress reactivity <sup>17-19</sup> are related to dropout. Despite this relationship, status quo treatment approaches do not account for physiological factors related to PTSD. <sup>20,21</sup> Due to these limitations, alternative interventions and treatment targets for PTSD are warranted.

**Mindfulness-Based Stress Reduction (MBSR) is a promising alternative.** <sup>1,22,23</sup> MBSR is a mindfulness-based intervention (MBI) and shows promise for treating PTSD in veterans. <sup>20,22,24-26</sup> MBSR improves PTSD symptoms and benefits physiological systems related to PTSD symptoms<sup>20</sup> such as the autonomic

nervous system.<sup>27</sup> Despite promising findings, <u>mechanisms by which MBSR may benefit PTSD are less</u> understood.<sup>28,29</sup>

Increased resilience may be the primary mechanism in MBSR for PTSD. Resilience is the ability to cope with, adapt to, or overcome exposure to stress.<sup>30</sup> Psychological resilience is conceptualized as a trait<sup>31-33</sup> or a teachable skill.<sup>34-37</sup> Psychological resilience is negatively associated with the likelihood of PTSD.<sup>38-40</sup> MBIs may reduce avoidance of trauma-related stressors, thereby increasing psychological resilience and reducing PTSD symptoms.<sup>41</sup> MBIs effectively increase psychological resilience high-stress groups,<sup>42,43</sup> and increased psychological resilience mediates improvements in stress disorders.<sup>44</sup>

Physiological resilience is another promising mechanism, and is defined as the capacity of a biological system to avoid shifting away from baseline (e.g., "reactivity") or to return to baseline (e.g., "recovery"). The sympathetic nervous system (SNS) has served as an indicator of physiological resilience among veterans. Physiologically, physiological resilience is indicated by the magnitude of peripheral vasoconstriction, and directly related to blood pressure (BP). BP has been conceptualized as an indicator of physiological resilience to negative health outcomes. Combat veterans with PTSD exhibit low physiological resilience via exaggerated BP reactivity to acute stress. The other research has found that trauma is predictive of lower physiological resilience. Ambstrates and resilience-based interventions reduce BP, improve physiological resilience, including among military personnel. Prior to conducting a fully-powered mechanistic RCT, central research methods such as intervention, stress induction, and physiological data collection must be validated.

**Feasibility and acceptability must be established.** Although some studies have conducted RCTs of MBSR among veterans with PTSD,<sup>23</sup> <u>feasibility and acceptability limitations remain</u>. A systematic review currently under review by the PI found that MBIs for PTSD showed an average attrition rate of 21.3%; <u>much higher than the general population.</u><sup>63</sup> The reason for this difference is unknown. A recent meta-analysis called for increased efforts to improve the feasibility and acceptability of MBIs.<sup>63</sup> Similarly, a recent review reported that data regarding adherence in MBSR (e.g. at-home meditation practice) is underreported in most studies.<sup>64</sup> <u>No studies have evaluated the feasibility and acceptability of these facets of MBSR among veterans with PTSD</u>. Further, no study has evaluated the feasibility and acceptability of a stressor task and concurrent physiological data collection in veterans. These aspects of feasibility require further study, as recent research has emphasized the need for stress induction tasks that are feasible and reproducible.<sup>65</sup> Given the novelty of these procedures in this population, and the potential impact of the PI's line of research among veterans underserved by status quo interventions, this KL2 application essential. To support this line of research, this KL2 will inform the resubmission of the PI's K23 proposal and forthcoming VA CDA.

**The long-term goal of this research** is to use mechanisms identified via a fully-powered mechanistic RCT funded by NIH K23 or VA CDA to optimize a resilience-based, trauma-informed MBI. In order to secure funding and conduct this mechanistic RCT, feasibility and acceptability of the stressor paradigm and concurrent physiological data collection, as well as the MBSR and randomization procedures must be established.

# 4) Study Design

The design of this study is a randomized controlled interventional study. All participants will complete three in-person lab visits, consisting of computerized questionnaires, physiological data recording, and completion of a stressor paradigm. Following completion of computerized questionnaires at the baseline visit, participants will be randomized at a 1:1 ratio using covariate adaptive randomization.

Participants will be randomized to receive Mindfulness-Based Stress Reduction (MBSR; active intervention condition) or Health and Wellness Education (HWE; control condition). Both interventions include 8 weekly in-person group sessions with an additional extended session after week 8.

# 5) Study Population

## a) Number of Subjects

This is a single center study. We will screen approximately 40 patients of which we expect to enroll 20 participants, all of whom will be veterans experiencing PTSD symptoms (PTSD symptoms will be confirmed during telephone screen). Therefore, 20 participants will sign the consent form and be included in this study.

#### b) Inclusion and Exclusion Criteria

Participants will be screened over phone to determine eligibility. Subjects will be aged 18-85 years. Subjects older than 85 years of age will be excluded due to their decreased ability to tolerate the experimental procedures because of potential cognitive decline and inability to sustain the attention needed for the Portland Arithmetic Stress Task (PAST), as well as the decreased ability to remain still during the intervention conditions due to musculoskeletal aches and pains and decreased flexibility frequently seen in aging.

| Inclusion criteria | Exclusion criteria |
|---|---|
| Adult (18-85 years) | Pregnancy |
| Military veteran | Severe untreated depression, cognitive impairment, or active suicidality* |
| Experiencing PTSD symptoms | Life-threatening or severely disabling medical conditions |
| Reading and speaking in English | Excessive use of alcohol, nicotine, or cannabis† |
| Be able to travel to OHSU for three two-hour lab visits, 8 weekly intervention sessions and one long extended session, and a two-hour focus group | |

<sup>\*</sup> Severe cognitive impairment will be determined by a score ≤ 20 on the Telephone Interview for Cognitive Status; active suicidality will be determined by endorsement of item 9 on the Patient Health Questionnaire.

If a participant does not consent, or is excluded for any other reason (e.g. screen-failed), data already collected (e.g., demographic; screening data) will be retained for the purpose of characterizing individuals who made contact, as well as collecting and presenting feasibility and acceptability data to the VEG at the conclusion of this study. The reason for not enrolling will be noted.

### c) Vulnerable Populations

No vulnerable populations will be recruited as part of this study.

<sup>†</sup> Alcohol use will be determined by a score ≥ 8 on the Alcohol Use Disorders Identification Test (AUDIT-C); excessive cannabis use will be determined by a score ≥ 7 on the Cannabis Abuse Screening Tool; excessive nicotine use will be determined by a score ≥8 on the Fagerstrom Nicotine Dependence Scale.

#### d) Setting

This is a single site study. All research activities, including interventions, will take place at OHSU with the exception of some recruitment procedures that will take place at the Portland VA (e.g., presenting study materials to clinics).

#### e) Recruitment Methods

A multi-dimensional recruitment strategy will be used to achieve target enrollment numbers. We will use OHSU approved recruitment tools such as Epic Reporting Workbench, Slicer Dicer, Research Data Warehouse (RDW), etc., to query OHSU electronic medical records. This study will use Epic MyChart® to recruit potential participants. Researchers will use OHSU approved search tools as mentioned above to identify potential study participants. Potential participants will be sent a MyChart® recruitment message asking them to participate. There is no risk of duplicate invitations as it is based on MyChart® accounts combined with Epic records and no duplication is possible.

Social media advertising and community outreach and snowball methods (e.g. word of mouth) will also be utilized as avenues for participant recruitment. With the approval of OHSU clinical providers and the OHSU IRB (with the support of the mentorship team), additional outreach will take place at OHSU using clinic lists of patients who have opted into research opportunities. Only passive recruitment will occur at the VAPORHCS. Specifically, VA clinic staff may provide approved flyer with OHSU study contact to any interested Veteran who in turn may reach out to the PI or study team with questions if interested. A potential participant may then call the study team at the number on the flyer to schedule a phone call to be screened for eligibility. Dr. Kaplan may also provide OHSU IRB approved flyer (including study contact information) to VAPORHCS clinicians not affiliated to the study team to provide to any veterans who elect not to initiate, or who discontinue traditional PTSD treatments (e.g., Cognitive Processing Therapy (CPT) or Prolonged Exposure (PE) prior to completion. In addition to these recruitment efforts through VAPORHCS and OHSU, flyers will be posted via online outlets such as Facebook and Craigslist, and recruitment materials will be distributed to veterans with the Multnomah County Veterans' Services. OHSU also hosts online search engines that allows potential participants to filter research participation opportunities based on certain criteria (e.g., compensation, time commitment). Dr. Kaplan will also present information about this study to veteran community resources, including Veterans of Foreign Wars (VFW) groups. Finally, Dr. Kaplan will engage in quarterly meetings with the Veterans Engagement Group (VEG) through VAPORHCS.

**Veterans Engagement Group (VEG).** The VEG is a 7-10 member group comprised entirely of veterans who are VAPORHCS patients, former employees, and clinicians. This group provides investigators with feedback throughout the research process. The VEG regularly assists researchers in maximizing their recruitment and retention efforts, as well as providing feedback on aspects such as qualitative data collection and analysis as presented in this proposal. Dr. Kaplan has been invited to attend regular VEG meetings in order to ensure the effectiveness of recruitment methods, and to discuss alternative strategies in the event of slow recruitment. VEG will not have access to any patient data or identifier. Dr. Kaplan may present aggregate recruitment/enrollment data to VEG in case there are problems and seek their advice to improve enrollment.

Interested veterans will contact the research team to be screened for eligibility and to be informed of the purpose and procedure of the study. They may reach out by seeing the online flyers on social media platforms or hearing about the study during clinic visits or being handed a flyer. As a secondary strategy, upon identification of Veterans through OHSU approved recruitment tools, we will send a letter via US postal service or an email to explain the study. A study team member's name and contact information will be provided in the letter so that the potential participant can call in to express interest or learn more about the study. Participants will also have the option to opt-out by calling or emailing the study team if

they wished not to be contacted. But if no response from the potential participant, the study team will call the Veterans who were sent the letters to discuss this study opportunity.

Participants will be screened for eligibility by phone using a standardized list of inclusionary and exclusionary questions (Initial phone contact). The study and the participants' right in research and compensation plan will be explained. Those who are eligible will be invited to a second phone screening which will be scheduled according to a time convenient to the participant. During the second screening visit, eligible participants will be asked some questions related to demographics and will be required to complete some survey questionnaires to gauge their quality of life, cognitive status, etc. (see table below). If the participant qualifies screening, someone from the team will contact the participant and inform them of their eligibility and next steps. Participant's name and contact information (phone number, mailing address, email address), age will be obtained to contact for the follow-up appointment and/or to initiate study participation. These identifiers will be kept in a separate database on the secured OHSU network drive or on OHSU acceptable cloud storage location.

Participants will be given modest financial compensation for attending study visits and intervention sessions: \$20 gift cards will be given at each study visit and post-intervention focus group interview (4 total), and \$5 will be added for each intervention session attended (9 total) for a total possible compensation amount of \$125 per participant. Compensation will be provided at the completion of each visit via ClinCard which will be reloaded following each visit. The amount compensated is comparable to the compensation provided in similar research studies and should adequately compensate for the time and travel involved without constituting undue pressure or influence on, or coercion of, the prospective research participants to volunteer for or continue participation in the research study.

#### **Consent Process**

Participants will be informed about their rights at the beginning of the telephone screening. The telephone screening confirms that adults are competent in reading and speaking English. It also confirms that adults are cognitively capable of consent through administration of the Telephone Interview for Cognitive Status. A HIPAA waiver of authorization (WOA) will allow for the collection of identifiable data before obtaining full consent in person. Information to be collected during screening are as follows:

#### **Screening Measures**

Abbreviated Posttraumatic Stress Disorder Checklist (PCL-6), depression (PHQ-9), suicidality (PHQ-9 item 9), substance use (Alcohol Use Disorders Identification Test; Cannabis Abuse Screening Tool; Fagerstrom Nicotine Dependence Scale), medical history, self-reported medication history, current mindfulness practice, historical mindfulness experience.

#### **Demographics**

Age, gender, sex, ethnicity, BMI, marital status, education, income, employment status, military branch, era of service, years enlisted.

Upon arrival at the research lab in Hatfield Research Center (HRC) for the first study visit, study personnel will review the study consent form with the participant and solicit questions. Once the subject verbally confirms understanding and interest in participation, they will be asked to sign consent forms and will be provided copies prior to leaving the HRC building. All research activities, including interventions, will take place at OHSU. Data collection and analysis will take place in the Oken Lab in OHSU's Hatfield Research Building, and interventions will take place at OHSU's Kohler Pavilion.

Subjects will be encouraged to ask questions throughout the duration of participation.

#### **Modifications to the Consent Process**

In this study, Veterans will primarily be recruited when they see a flyer and contact the study team. The PI will not be accessing the VA electronic medical record to identify a potential patient. Once a potential participant reaches out to the PI and study from the contact information provided in the flyer, the PI or a delegated study team member will review the initial phone script to understand if the participant meets eligibility and shows interest in participation. If the veteran is interested, the study team will call the participant at an agreed upon time to conduct screening procedures over phone. If the participant is eligible, the participant will be invited to sign the OHSU informed consent form prior to randomizing to the study intervention (MBSR or HWE).

We believe that requesting the participant to sign the consent form after screening will not adversely affect the patient as we will have a waiver to store this information in the secure network drive at OHSU. We have carefully selected the data elements as the minimum necessary in order to identify and recruit potentially eligible Veterans into this study without placing undue burden on the veterans. This is a minimal-risk study. Patients can avoid an unnecessary visit at OHSU to sign the consent form if they are ultimately determined to be not eligible after screening.

## Non-English Speaking Subjects

English language reading and speaking are inclusion criteria for this study. Certain elements of the protocol such as the stressor task (Portland Arithmetic Stress Task) are not validated in other languages and would therefore not be able to be applied uniformly.

#### **Assent of Children and Parent Permission**

This is a study on Veterans so children will not be included.

#### Adults Unable to Consent/Decisionally Impaired

No decisionally-impaired adults will be recruited, and cognitive status will be determined during the phone screen.

### 6) Procedures

Aim 1 – Quantitative data: Recruitment and retention rates will be collected, compared between conditions, and evaluated in relation to previous research on MBSR recruitment and attrition. Correlations between rates of home practice completion (e.g., self-guided meditation practice) and attrition rates per condition will be examined for relationships. This quantitative data will be used to guide focus group prompt development.

Aims 1&2 – Qualitative data: Focus groups will be conducted in accordance with guidelines for maximizing impact of qualitative research in feasibility studies. <sup>66</sup> Broad topics will cover: 1) intervention content, 2) trial design and process (including stress induction and concurrent physiological data collection), 3) outcomes, and 4) measures. These discussion topics will be tailored to fit combat veterans with PTSD symptoms via consultation with the Veteran's Engagement Group (VEG; see *Human Subject Considerations* for a description of the VEG; see also Matsumoto LOS). A thematic analysis approach<sup>67</sup> will explore participant experiences to understand feasibility, acceptability, and impact of assessments, protocol, and interventions. Analysis process will consist of: 1) familiarization, 2) initial coding, 3) creating themes, 4) reviewing themes, 5) defining and naming themes, and 6) data interpretation. The PI will work with Dr. Christopher (co-mentor) who has experience conducting thematic analysis of qualitative data in feasibility studies, and a trained RA to independently review focus group data. Emerging themes will help develop a coding scheme that the team will apply independently the finalized code structure. The team will meet regularly to review coding and discrepancies to ensure inter-rater reliability.

**Aim 2 – Physiological data:** We will assess feasibility and effectiveness of stress induction by analyzing change in blood pressure (BP) between baseline and a cognitive stressor (see *Stress induction paradigm* 

section below). BP will be collected via Caretaker Medical VitalStream™ device, which accurately and wirelessly measures vital signs. The VitalStream™ uses an automated readout inflatable finger cuff and is connected via Bluetooth to a tablet. Within-participants baseline-to-stressor task t-tests will evaluate feasibility of stress induction. Significant increases in BP from baseline to stressor will constitute effective stress induction. Quantitative analyses will be conducted in SPSS v.28,<sup>68</sup> and qualitative will be conducted in NVivo.<sup>69</sup>

Stress induction: **1. Baseline:** The Simple Reaction Task (SRT) will serve as a baseline for the stressor task. Participants press a key each time a number appears on the screen. The SRT has been used as a baseline for cognitive stressors in prior Oken lab studies; **2. Stress induction:** The Portland Arithmetic Stress Task (PAST)<sup>70</sup> is a cognitive stressor comprised of arithmetic problems titrated in difficulty. It has an adaptive failure algorithm, maintaining an error rate of ~40%. It has been shown to induce physiological stress across groups. <sup>70-72</sup>

Aim 3 – Quantitative data will be collected on paper and entered in REDCap by a study team member on an Oken lab computer and in-person clinical interview (i.e., Clinician-Administered PTSD Scale for DSM-5 [CAPS-5]). Using this data, we will examine sensitivity and responsiveness to change of outcomes. This Aim will be conducted in accordance with best practice guidelines, 73,74 CONSORT recommendations,<sup>75</sup> and previous research.<sup>76,77</sup> Sensitivity in both groups will be analyzed via relative efficiency; dividing the F-statistic for each physiological (systolic and diastolic BP) and self-report (psychological resilience and PTSD symptoms) by the largest F-statistic among outcomes (see Table below for measures). 77,78 This process will clarify which outcomes are most sensitive to MBSR. To generate F-statistics for relative efficiency, we will conduct repeated measures ANOVAs for each outcome in both groups. This statistical approach focuses on the degree to which measures are sensitive, not whether change is significant. Responsiveness to change over time will be assessed in the MBSR group for physiological and self-report outcomes by: 1) calculating and comparing standardized mean response by subtracting baseline mean response from post-intervention mean response, and dividing by standard deviation of change 14,79,80 and 2) examining zero-order correlations between a global impression of change measure (post-intervention) and change scores (baseline to postintervention) for self-report outcomes.<sup>81-83</sup>

Primary measures to be collected are listed below:

| Method | Variable | Measurement Tool | Timepoints |
|---|---|---|---|
| Paper>REDCap | Psychological resilience | Brief Resilience Scale (BRS) | Pre, mid, post |
| Paper>REDCap | PTSD symptoms | PTSD Symptoms Checklist for DSM-5 (PCL-5) | Pre, mid, post |
| Paper>REDCap | Mindfulness | Five Facet Mindfulness Questionnaire (FFMQ-15) | Pre, mid, post |
| Paper>REDCap | Perceived stress | Perceived Stress Scale (PSS-10) | Pre, mid, post |
| Paper>REDCap | Loneliness | UCLA Loneliness Scale | Pre, mid, post |
| Paper>REDCap | Distress | Distress tolerance scale | Pre, mid, post |
| Clinical interview | PTSD symptoms | Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Pre, mid, post |
| CareTaker™ | Physiological resilience | Blood pressure (BP) | Pre, mid, post |

Stress induction: **1. Baseline:** The Simple Reaction Task (SRT) will serve as a baseline for the stressor task. Participants press a key each time a number appears on the screen. The SRT has been used as a baseline for cognitive stressors in prior Oken lab studies; **2. Stress induction:** The Portland Arithmetic Stress Task (PAST)<sup>70</sup> is a cognitive stressor comprised of arithmetic problems titrated in difficulty. It has an adaptive failure algorithm, maintaining an error rate of ~40%. It has been shown to induce physiological stress across groups. <sup>70-72</sup>

#### Interventions:

**Mindfulness-Based Stress Reduction** consists of weekly two-hour sessions for eight weeks, and a 7 hour retreat after Lab visit 3/week 8. The MBSR intervention will be facilitated by an experienced and

certified MBSR teacher. MBSR curriculum strongly encourages completion of home practice assignments (~30 minutes daily) to help integration of concepts into daily life. Participants will receive audio CDs and a DVD to help guide home practice.

Health and Wellness Education (HWE) Intervention is a didactic-based group intervention designed as an active comparator for randomized-controlled trials of MBSR. HWE provides instruction to participants regarding improving their emotional and physical health. In contrast to MBSR, there are no attempts to train participants' breathing, movement, or meditation habits or practices. HWE is administered in 8 weekly 2.5-hour classes with home practice to be completed between sessions (matched to MBSR for amount and effort). HWE also features one extended 7hour retreat, similar to MBSR. <sup>84</sup> Dr. Autumn Gallegos (consultant) has conducted trials of MBSR among veterans with PTSD using a control group based on similar materials, and will provide mentorship to the PI in administering the control intervention. Dr. Kaplan and a trained RA will facilitate HWE.

CareTaker VitalStream™. The CareTaker VitalStream™ is comprised of a lightweight wrist pack attached via Velcro, which is connected via thin tube to a small Velcro finger cuff that contains a low-pressure sensor. All materials used in the VitalStream™ are medical grade. VitalStream™ measures continuous pulse pressure waveforms for processing via Pulse Decomposition Analysis™ (PDA™). The PDA™ technology includes algorithms to calculate and continuously monitor hemodynamic-related parameters by analyzing reflective pulsewave morphology within the arterial system. The VitalStream™ allows for secure wireless monitoring via a real-time mobile application, or remote monitoring via a Cloud Portal. For the purposes of the study, we will monitor participant data via mobile application on an encrypted Android tablet in a room adjacent to the testing room during the laboratory stressor task. Dr. Kaplan (PI) designed and executed a pilot RCT using a previous version of CareTaker. Through this study Dr. Kaplan gained familiarity with the equipment and software, and developed relationships with key CareTaker Medical personnel.

**Blood pressure.** The VitalStream™ measures and records systolic, diastolic, and mean arterial pressure (MAP) using FDA-approved PDA™ technology. These algorithms have been validated in comparison to invasive central aortic measurement.

**Heart rate.** The VitalStream<sup>™</sup> measures heart rate via low-pressure finger sensor, with accuracy validated in comparison to 3-lead ECG measurement.

**Respiration rate.** The VitalStream<sup>™</sup> accurately measures respiration rate (breaths per minute) non-invasively by extrapolating pulsewave morphology via PDA<sup>™</sup>. The VitalStream<sup>™</sup> calculates respiration rate in this fashion with equivalent accuracy to ECG-derived respiration using a 3-lead ECG electrode.

Potential participants will be sent a MyChart recruitment invitation and a follow-up (as applicable) via an email notification, as below, with the Subject "New Research Study" instructing them to log into MyChart to learn more and respond. The text of this invitation is included in the eIRB submission. The link in the MyChart invitation will take the potential participant to their MyChart homepage with a link to a description of the study. Potential participants will express interest or decline by pressing the associated buttons in MyChart, or they will not respond. If the potential participant indicates interest, they are automatically associated to the study in Epic with a status of "interested;" the study remains listed on the patient's Research Studies page in MyChart, and the study team immediately receives an in-basket notification in Epic so that they can follow up with the patient. If the patient clicks "No, Thank You" this study will no longer appear on their Research Studies page in MyChart, and the patient is automatically associated to the study in Epic with a status of "declined." When the participant expresses interest, the study team will call the participant to schedule the initial phone call for an initial review of eligibility and a second screening phone call before the participant is enrolled on study. Details of the initial and second phone call are included under "recruitment methods" section.

Please see below for a description of the study schedule. All survey data will be captured in paper surveys from study participants and will be directly entered in the REDCap database by a study team member.

#### Study Schedule:

| Visits | Initial<br>phone<br>call 1 | Screening phone call | Lab visit<br>1 | Wk<br>1 <sup>e</sup> | Wk<br>2 | Wk<br>3 | Wk<br>4 | Wk5/<br>Lab<br>visit 2 | Wk<br>6 | Wk<br>7 | Wk8/<br>Lab<br>visit 3 | Retreat | Post-<br>interventi<br>on Wk9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study overview and eligibility review | Х | | | | | | | | | | | | |
| Screening questionnaires <sup>a</sup> | | Х | | | | | | | | | | | |
| Demographics <sup>b</sup> | | Х | | | | | | | | | | | |
| Informed consent | | | Х | | | | | | | | | | |
| MBSR/HWE <sup>d</sup> intervention | | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Study Visit<br>Questionnaires <sup>c</sup> | | | Х | | | | | Х | | | Х | | |
| Clinical<br>interview<br>(Clinician<br>administered<br>PTSD scale for<br>DSM-5 (CAPS-5) | | | Х | | | | | Х | | | Х | | |
| CareTaker VitalStream™ (physiologic data collection, BP) | | | Х | | | | | Х | | | X | | |
| Lab Stressor | | | X | | | | | Χ | | | Χ | | |
| Focus group<br>Qualitative<br>interview | | | | | | | | | | | | | Х |
| Approximate total time | 15 mins | 30 mins | 120 mins | 150<br>mins | 150<br>mins | 150<br>mins | 150<br>mins | 270<br>mins | 150<br>mins | 150 | 270<br>mins | 7 hours | 120 mins |

- a. Screening measures will include: PTSD (PCL-5), depression (PROMIS), suicidality (PHQ-9), substance abuse (Alcohol Use Disorders Identification Test, Cannabis Abuse Screening Tool, Fagerstrom Nicotine Dependence Scale) in addition to review of eligibility
- b. Demographic information includes age, gender, sex, ethnicity, BMI, marital status, education, income, employment status, military branch, era of service, years enlisted. Medical and medication history, current and historical mindfulness experience are captured during screening
- c. Questionnaires include Brief Resilience Scale, PTSD Symptoms Checklist for DSM-5 (PCL-5,6), UCLA Loneliness Scale, CAPS-5, Five Facet Mindfulness Questionnaire (FFMQ-15), Perceived Stress Scale (PCL-10), Distress tolerance scale (DTS)
- d. Participants are randomized at visit 1 to either MBSR or HWE. All participants have 30-minute practice assignments to be carried out every day at home.
- e. Week 1 of the interventions will occur within one week of completing Lab Visit 1 for all participants.

Participants may be withdrawn from this study without their consent in order to protect them from excessive risk (e.g., if they demonstrate unsafe elevated blood pressure), or in order to maintain the integrity of the study and data (e.g., a participant is not following study procedures and/or may be deliberately providing false information).

#### 7) Data

#### **Handling of Data**

Data collected will include computer-based and physiological recordings listed above, as well as demographic data such as age and gender. Data will also include health status information, such as

medical conditions and prescription medications for use in determining eligibility. All data will be stored on a restricted OHSU network drive in a limited access folder or in a REDCap database, and the study PI and designee will be responsible for storage and transmission of the data. Following this study, all data will be transferred and stored indefinitely in repository IRB #7436. No specimens will be collected as part of this study.

#### a) Sharing of Results with Subjects

Participants will be given the opportunity to view their heart rate and blood pressure when it is taken in the lab during the baseline condition, unless they would prefer not to. Participants will not be shown their physiological data during the stressor condition due to the expected increases resulting from cognitive stress. Besides this, participants will not have access to any other data collected as a part of this study. If participants demonstrate pathological blood pressure during the course of the study, they will be notified and referred to their PCP and/or urgent care. If blood pressure reaches hypertensive crisis (180/110) the participant will be referred immediately to the emergency department. No data will be used for clinically decision-making, nor will it be entered into participants' medical records. Referrals will be made based on generic critical blood pressure values only.

#### b) Data and Specimen Banking

If data or specimens will be banked in a repository for future use as part of this protocol submission, describe here (or in a separate repository protocol document) where they will be stored, how long they will be stored, how they may be accessed, and who will have access to the specimens. Describe the procedures to release data or specimens, including: the process to request a release, approvals required for release, who can obtain data or specimens, and the data to be provided with specimens.

Data will be sent to a repository maintained separately from this study. They will be stored indefinitely in repository IRB #7436. Participants will be requested to consent to sharing data in the repository which will be optional. The repository investigator and members of the Oken Cognitive Neuroscience Laboratory are allowed to access the data and will have requisite HIPAA and other trainings. Please see repository protocol for details related to that study.

## 8) Data Analysis

Quantitative data:

Recruitment and retention rates will be collected, compared between conditions, and evaluated in relation to previous research on MBSR recruitment and attrition. Correlations between rates of home practice completion (e.g., self-guided meditation practice) and attrition rates per condition will be examined for relationships.

Within-participants baseline-to-stressor task t-tests will evaluate feasibility of physiological stress induction. Significant increases in BP from baseline to stressor will constitute effective stress induction.

<u>Sensitivity</u> in both groups will be analyzed via relative efficiency; dividing the F-statistic for each physiological (systolic and diastolic BP) and self-report (psychological resilience and PTSD symptoms) by the largest F-statistic among outcomes (see Table above for measures). This process will clarify which outcomes are most sensitive to MBSR. To generate F-statistics for relative efficiency, we will conduct repeated measures ANOVAs for each outcome in both groups. This statistical approach focuses on the degree to which measures are sensitive, not whether change is significant. Responsiveness to change over time will be assessed in the MBSR group for physiological and self-report outcomes by: 1) calculating and comparing standardized mean response by subtracting baseline mean response from post-intervention mean response, and dividing by standard deviation of change T4,79,80 and 2) examining zero-order correlations between

a global impression of change measure (post-intervention) and change scores (baseline to post-intervention) for self-report outcomes.<sup>81-83</sup>

#### Qualitative data:

A thematic analysis approach<sup>67</sup> to qualitative data will explore participant experiences to understand feasibility, acceptability, and impact of assessments, protocol, and interventions. Analysis process will consist of: 1) familiarization, 2) initial coding, 3) creating themes, 4) reviewing themes, 5) defining and naming themes, and 6) data interpretation.

# 9) Privacy, Confidentiality and Data Security

Standard institutional practices will be followed as described in the OHSU Information Security Directives (http://www.ohsu.edu/xd/about/services/integrity/policies/ips-policies-info-sec-directiv.cfm#results) to maintain the confidentiality and security of data collected in this study. Study staff will be trained with regard to these procedures. Any staff that will be involved in these research activities will have completed the requisite Human Subject Protection Training as required by the IRB prior to engagement. Documentation of training will be held on secure password protected computers at OHSU. Prior to implementation of any protocol changes, amendments will be submitted to the OHSU Institutional Review Board for approval. Dr. Kaplan will be responsible for continuous data and safety monitoring of all participants, and discussion of any data or safety monitoring concerns will be a routine topic of mentorship and consultation meetings. In the event there are AEs/SAEs that require medical intervention, Dr. Oken, a board-certified neurologist, will be available to review events and refer them as needed.

Paper files will be stored in locked filing cabinets in restricted access offices at OHSU and will not leave the Oken lab facility. Electronic data is stored on restricted drives on the OHSU network, on OHSU approved cloud location and on encrypted computers. Electronic data will also be stored in a custom database housed on an OHSU secure server. Access to data is restricted to study personnel. Access to data requires OHSU ID/password authentication.

Upon enrollment, participants will be assigned a code that will be used instead of their name, medical record number or other personally identifying information. Electronic files for data analysis will contain only the subject code. Codes will not contain any part of the 18 HIPAA identifiers (initials, DOB, MRN) The key associating the codes and the participants personally identifying information will be restricted to the PI and study staff. The key will be kept secure on a restricted OHSU network drive in a limited access folder.

BP will be collected via Caretaker Medical VitalStream™ device, which accurately and wirelessly measures vital signs. The VitalStream™ uses an automated readout inflatable finger cuff and is connected via Bluetooth to a tablet. The CareTaker™ is completely wireless, and will relay data via Bluetooth connectivity to a tablet. It allows for secure wireless monitoring via a real-time mobile application, or remote monitoring via a Cloud Portal. For the purposes of the study, we will monitor participant data via mobile application on an encrypted Android tablet in a room adjacent to the testing room during the laboratory stressor task. There is no storage, processing or transmission of any PHI or HIPAA identifiers through VitalStream. It does not connect to OHSU network, but is transmitted via Bluetooth to an encrypted tablet.

At the completion of the study, if patients consent to sharing data in the repository, their data will be released to repository IRB #7436. See repository protocol for details about requesting, releasing, and labeling data.

# 10) Risks and Benefits

## a) Risks to Subjects

The risk in participating in the present study is low. Participants may feel distress when reporting their PTSD symptoms or identifying their index trauma (i.e., the most salient trauma connected to their PTSD symptoms) as part of the administration of the Clinician-Administered PTSD Scale (CAPS-5). Participants may also feel discomfort or embarrassment when discussing their general experiences during the intervention conditions. They may also feel stress or frustration when completing the laboratory stressor paradigm. Participants have the right to withdraw, and may attend intervention groups and not actively participate, or may not complete MBSR home practice between sessions.

There is no discomfort associated with the collection of physiological data. The CareTaker™ device using a Velcro finger cuff attached with similar tightness to an arm cuff blood pressure monitor. A thin clear tube connects the finger cuff to a small wrist pack that houses the electronic components of the device. The CareTaker™ is completely wireless, and will relay data via Bluetooth connectivity to a tablet.

One of the potential risks of participation breach of confidentiality. It is possible that, if someone inadvertently obtained data, this could result in harm to research participants, with legal, financial, or emotional implications of the affected Veterans. We will take all possible measures to protect the security and integrity of personal health information.

#### b) Potential Benefits to Subjects

Veterans may find it rewarding to engage in group-based interventions in which they are encouraged to share their experiences with other veterans with similar struggles related to PTSD symptoms. They may similarly appreciate being able to share their perspectives regarding their ability and strategies for coping with symptoms. Participants may also experience reduction in symptoms of PTSD, depression, and anxiety as a result of participating in the MBSR condition.

#### REFERENCES

1. Boyd JE, Lanius RA, McKinnon MC. Mindfulness-based treatments for posttraumatic stress disorder: a review of the treatment literature and neurobiological evidence. J Psychiatry Neurosci 2018;43(1):7-25. (In eng). DOI: 10.1503/jpn.170021.

- 2. Hilton L, Maher AR, Colaiaco B, et al. Meditation for posttraumatic stress: Systematic review and metaanalysis. Psychological trauma: theory, research, practice and policy 2017;9(4):453-460. (In eng). DOI: 10.1037/tra0000180.
- 3. Banks K, Newman E, Saleem J. An Overview of the Research on Mindfulness-Based Interventions for Treating Symptoms of Posttraumatic Stress Disorder: A Systematic Review. Journal of clinical psychology 2015;71(10):935-63. (In eng). DOI: 10.1002/jclp.22200.
- 4. Boscarino JA. A prospective study of PTSD and early-age heart disease mortality among Vietnam veterans: implications for surveillance and prevention. Psychosomatic medicine 2008;70(6):668-676. (In eng). DOI: 10.1097/PSY.0b013e31817bccaf.
- 5. Tanielian T, Jaycox LH, Schell TL, et al. Invisible Wounds: Mental Health and Cognitive Care Needs of America's Returning Veterans: RAND Corporation, 2008.
- 6. Davidson JR. Pharmacologic treatment of acute and chronic stress following trauma: 2006. The Journal of clinical psychiatry 2006;67 Suppl 2:34-9. (In eng).
- 7. Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. The American journal of psychiatry 2005;162(2):214-27. (In eng). DOI: 10.1176/appi.ajp.162.2.214.
- 8. Kim SH, Schneider SM, Kravitz L, Mermier C, Burge MR. Mind-body practices for posttraumatic stress disorder. Journal of investigative medicine: the official publication of the American Federation for Clinical Research 2013;61(5):827-34. (In eng). DOI: 10.2310/JIM.0b013e3182906862.
- 9. VA/DOD Clinical Practice Guideline for the Management of Posttraumatic Stress Disorder and Acute Stress Disorder: Clinician Summary. FOCUS 2018;16(4):430-448. DOI: 10.1176/appi.focus.16408.
- 10. Asmundson GJ, Thorisdottir AS, Roden-Foreman JW, et al. A meta-analytic review of cognitive processing therapy for adults with posttraumatic stress disorder. Cognitive Behaviour Therapy 2019;48(1):1-14.
- 11. Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clinical psychology review 2010;30(6):635-641.
- 12. Bisson JI, Ehlers A, Matthews R, Pilling S, Richards D, Turner S. Psychological treatments for chronic post-traumatic stress disorder: Systematic review and meta-analysis. The British journal of psychiatry 2007;190(2):97-104.
- 13. Grunert BK, Weis JM, Smucker MR, Christianson HF. Imagery rescripting and reprocessing therapy after failed prolonged exposure for post-traumatic stress disorder following industrial injury. J Behav Ther Exp Psychiatry 2007;38(4):317-28. (In eng). DOI: 10.1016/j.jbtep.2007.10.005.
- 14. Kehle-Forbes SM, Meis LA, Spoont MR, Polusny MA. Treatment initiation and dropout from prolonged exposure and cognitive processing therapy in a VA outpatient clinic. Psychological trauma: theory, research, practice and policy 2016;8(1):107-114. (In eng). DOI: 10.1037/tra0000065.
- 15. Schottenbauer MA, Glass CR, Arnkoff DB, Tendick V, Gray SH. Nonresponse and dropout rates in outcome studies on PTSD: review and methodological considerations. Psychiatry 2008;71(2):134-68. (In eng). DOI: 10.1521/psyc.2008.71.2.134.
- 16. Goetter EM, Bui E, Ojserkis RA, Zakarian RJ, Brendel RW, Simon NM. A Systematic Review of Dropout From Psychotherapy for Posttraumatic Stress Disorder Among Iraq and Afghanistan Combat Veterans. J Trauma Stress 2015;28(5):401-9. (In eng). DOI: 10.1002/jts.22038.
- 17. Zayfert C, DeViva JC, Becker CB, Pike JL, Gillock KL, Hayes SA. Exposure Utilization and Completion of Cognitive Behavioral Therapy for PTSD in a "Real World" Clinical Practice. Journal of Traumatic Stress 2005;18(6):637-645. DOI: 10.1002/jts.20072.
- 18. Garcia HA, Kelley LP, Rentz TO, Lee S. Pretreatment predictors of dropout from cognitive behavioral therapy for PTSD in Iraq and Afghanistan war veterans. Psychological Services 2011;8(1):1-11. DOI: 10.1037/a0022705.
- 19. Alpert E, Hayes AM, Barnes JB, Sloan DM. Predictors of dropout in cognitive processing therapy for PTSD: An examination of trauma narrative content. Behavior Therapy 2020;51(5):774-788.

Protocol version 2.4

- 20. Bremner JD, Mishra S, Campanella C, et al. A Pilot Study of the Effects of Mindfulness-Based Stress Reduction on Post-traumatic Stress Disorder Symptoms and Brain Response to Traumatic Reminders of Combat in Operation Enduring Freedom/Operation Iraqi Freedom Combat Veterans with Post-traumatic Stress Disorder. Front Psychiatry 2017;8:157. (In eng). DOI: 10.3389/fpsyt.2017.00157.
- 21. Shepherd L, Wild J. Emotion regulation, physiological arousal and PTSD symptoms in trauma-exposed individuals. Journal of Behavior Therapy and Experimental Psychiatry 2014;45(3):360-367. DOI: https://doi.org/10.1016/j.jbtep.2014.03.002.
- 22. Kearney DJ, Simpson TL, Malte CA, Felleman B, Martinez ME, Hunt SC. Mindfulness-based Stress Reduction in Addition to Usual Care Is Associated with Improvements in Pain, Fatigue, and Cognitive Failures Among Veterans with Gulf War Illness. Am J Med 2016;129(2):204-14. (In eng). DOI: 10.1016/j.amjmed.2015.09.015.
- 23. Taylor J, McLean L, Korner A, Stratton E, Glozier N. Mindfulness and yoga for psychological trauma: systematic review and meta-analysis. J Trauma Dissociation 2020:1-38. (In eng). DOI: 10.1080/15299732.2020.1760167.
- 24. Davis LL, Whetsell C, Hamner MB, et al. A Multisite Randomized Controlled Trial of Mindfulness-Based Stress Reduction in the Treatment of Posttraumatic Stress Disorder. Psychiatric Research and Clinical Practice 2019;1(2):39-48. (https://doi.org/10.1176/appi.prcp.20180002). DOI: https://doi.org/10.1176/appi.prcp.20180002.
- 25. Kearney DJ, McDermott K, Malte C, Martinez M, Simpson TL. Effects of participation in a mindfulness program for veterans with posttraumatic stress disorder: a randomized controlled pilot study. Journal of clinical psychology 2013;69(1):14-27. (In eng). DOI: 10.1002/jclp.21911.
- 26. Polusny MA, Erbes CR, Thuras P, et al. Mindfulness-Based Stress Reduction for Posttraumatic Stress Disorder Among Veterans: A Randomized Clinical Trial. Jama 2015;314(5):456-65. (In eng). DOI: 10.1001/jama.2015.8361.
- 27. Nijjar PS, Puppala VK, Dickinson O, et al. Modulation of the autonomic nervous system assessed through heart rate variability by a mindfulness based stress reduction program. International journal of cardiology 2014;177(2):557-559.
- 28. Schure MB, Simpson TL, Martinez M, Sayre G, Kearney DJ. Mindfulness-Based Processes of Healing for Veterans with Post-Traumatic Stress Disorder. Journal of alternative and complementary medicine (New York, NY) 2018;24(11):1063-1068. (In eng). DOI: 10.1089/acm.2017.0404.
- 29. Williston SK, Grossman D, Mori DL, Niles BL. Mindfulness interventions in the treatment of posttraumatic stress disorder. Professional Psychology: Research and Practice 2021;52(1):46-57. DOI: 10.1037/pro0000363.
- 30. Meredith LS, Sherbourne CD, Gaillot SJ, et al. Promoting Psychological Resilience in the U.S. Military. Rand health quarterly 2011;1(2):2. (In eng).
- 31. Tugade M, Fredrickson B, Barret L. Psychological resilience and positive emotional granularity: Examining the benefits of positive emotions on coping and health. Journal of Personality 2004;72(6):1161-1190.
- 32. Block J, Kremen A. IQ and ego-resiliency: Conceptual and empirical connections and separateness. Journal of Personality and Social Psychology 1996(70):349-361.
- Tugade M, Fredrickson B. Positive emotions and emotional intelligence. In: Barret L, Salovey P, eds. The Wisdom of Feelings. New York: Guilford; 2002:319-340.
- 34. Agaibi C, JP W. Trauma, PTSD, and resilience. Trauma, Violence, & Abuse 2005;6(3):195-216.
- 35. Masten A, Best K, Garmezy N. Resilience and development: Contributions from the study of children who overcame adversity. Development and Psychopathology 1990(2):425-444.
- 36. Reynolds A. Resilience among black urban youth: Prevalence, intervention effects, and mechanisms of influence. American Journal of Orthopsychiatry 1998(68):84-100.
- 37. Tarter R, Vanyukov M. Re-visiting the validity of the construct of resilience. In: Glantz M, Johnson J, eds. Resiliency and development: Positive life adaptations. New York: Plenum; 1999:85-100.

Protocol version 2.4

- 38. Wrenn GL, Wingo AP, Moore R, et al. The effect of resilience on posttraumatic stress disorder in traumaexposed inner-city primary care patients. J Natl Med Assoc 2011;103(7):560-6. (In eng). DOI: 10.1016/s0027-9684(15)30381-3.
- 39. Green KT, Calhoun PS, Dennis MF, Beckham JC. Exploration of the resilience construct in posttraumatic stress disorder severity and functional correlates in military combat veterans who have served since September 11, 2001. The Journal of clinical psychiatry 2010;71(7):823-30. (In eng). DOI: 10.4088/JCP.09m05780blu.
- 40. Pietrzak RH, Johnson DC, Goldstein MB, et al. Psychosocial buffers of traumatic stress, depressive symptoms, and psychosocial difficulties in veterans of Operations Enduring Freedom and Iraqi Freedom: The role of resilience, unit support, and postdeployment social support. Journal of Affective Disorders;120(1):188-192. DOI: 10.1016/j.jad.2009.04.015.
- 41. Thompson RW, Arnkoff DB, Glass CR. Conceptualizing Mindfulness and Acceptance as Components of Psychological Resilience to Trauma. Trauma, Violence, & Abuse 2011;12(4):220-235. DOI: 10.1177/1524838011416375.
- 42. Christopher MS, Hunsinger M, Goerling LRJ, et al. Mindfulness-based resilience training to reduce health risk, stress reactivity, and aggression among law enforcement officers: A feasibility and preliminary efficacy trial. Psychiatry research 2018;264:104-115. (In eng). DOI: 10.1016/j.psychres.2018.03.059.
- 43. Christopher M, Goerling R, Rogers B, et al. A Pilot Study Evaluating the Effectiveness of a Mindfulness-Based Intervention on Cortisol Awakening Response and Health Outcomes among Law Enforcement Officers. J Police Crim Psych 2015:1-14. (In English). DOI: 10.1007/s11896-015-9161-x.
- 44. Kaplan JB, Bergman AL, Hunsinger M, Bowen S, Christopher M. Resilience mediates the relationship between mindfulness training and burnout among first responders. 2016.
- Oken BS, Chamine I, Wakeland W. A systems approach to stress, stressors and resilience in humans. Behavioural Brain Research 2015;282:144-154. DOI: <a href="http://dx.doi.org/10.1016/j.bbr.2014.12.047">http://dx.doi.org/10.1016/j.bbr.2014.12.047</a>.
- 46. Beckner ME, Main L, Tait J, Martin BJ, Conkright WR, Nindl BC. CIRCULATING BIOMARKERS ASSOCIATED WITH PERFORMANCE AND RESILIENCE DURING MILITARY OPERATIONAL STRESS: Biomarkers associated with resilience in military operational stress. European journal of sport science 2021(just-accepted):1-33.
- 47. Baker DG, Nash WP, Litz BT, et al. Predictors of risk and resilience for posttraumatic stress disorder among ground combat Marines: methods of the Marine Resiliency Study. Prev Chronic Dis 2012;9:E97. (In eng). DOI: 10.5888/pcd9.110134.
- 48. Ortega M, Saavedra S. Resilience: physiological assembly and phychosocial factors. Procedia-social and behavioral sciences 2014;132:447-453.
- 49. WESSELING KH, SETTELS JJ, HOEVEN GMVD, NIJBOER JA, BUTIJN MW, DORLAS JC. Effects of peripheral vasoconstriction on the measurement of blood pressure in a finger. Cardiovascular research 1985;19(3):139-145.
- 50. Sabayan B, Oleksik AM, Maier AB, et al. High blood pressure and resilience to physical and cognitive decline in the oldest old: the Leiden 85-plus Study. J Am Geriatr Soc 2012;60(11):2014-9. (In eng). DOI: 10.1111/j.1532-5415.2012.04203.x.
- 51. Buckley TC, Holohan D, Greif JL, Bedard M, Suvak M. Twenty-Four-Hour Ambulatory Assessment of Heart Rate and Blood Pressure in Chronic PTSD and Non-PTSD Veterans. Journal of Traumatic Stress 2004;17(2):163-171. DOI: 10.1023/B:JOTS.0000022623.01190.f0.
- 52. Edmondson D, Sumner JA, Kronish IM, Burg MM, Oyesiku L, Schwartz JE. The Association of Posttraumatic Stress Disorder With Clinic and Ambulatory Blood Pressure in Healthy Adults. Psychosomatic medicine 2018;80(1):55-61. (In eng). DOI: 10.1097/PSY.0000000000000523.
- 53. Szabo YZ, Fernandez-Botran R, Newton TL. Cumulative trauma, emotion reactivity and salivary cytokine levels following acute stress in healthy women. Anxiety, Stress, & Coping 2019;32(1):82-94. DOI: 10.1080/10615806.2018.1524377.

01.03.2024 Page 15 of 17 Template Revised: 6.15.2015

- 54. Solano López AL. Effectiveness of the Mindfulness-Based Stress Reduction Program on Blood Pressure: A Systematic Review of Literature. Worldviews on Evidence-Based Nursing 2018;15(5):344-352. (https://doi.org/10.1111/wvn.12319). DOI: https://doi.org/10.1111/wvn.12319.
- 55. Momeni J, Omidi A, Raygan F, Akbari H. The effects of mindfulness-based stress reduction on cardiac patients' blood pressure, perceived stress, and anger: a single-blind randomized controlled trial. Journal of the American Society of Hypertension 2016;10(10):763-771. DOI: https://doi.org/10.1016/j.jash.2016.07.007.
- 56. Campbell TS, Labelle LE, Bacon SL, Faris P, Carlson LE. Impact of Mindfulness-Based Stress Reduction (MBSR) on attention, rumination and resting blood pressure in women with cancer: A waitlist-controlled study. Journal of Behavioral Medicine 2012;35(3):262-271. DOI: 10.1007/s10865-011-9357-1.
- 57. Nyklíček I, Mommersteeg PMC, Van Beugen S, Ramakers C, Van Boxtel GJ. Mindfulness-based stress reduction and physiological activity during acute stress: A randomized controlled trial. Health Psychology 2013;32(10):1110-1113. DOI: 10.1037/a0032200.
- 58. Intarakamhang U, Macaskill A, Prasittichok P. Mindfulness interventions reduce blood pressure in patients with non-communicable diseases: A systematic review and meta-analysis. Heliyon 2020;6(4):e03834. DOI: <a href="https://doi.org/10.1016/j.heliyon.2020.e03834">https://doi.org/10.1016/j.heliyon.2020.e03834</a>.
- 59. Steinhardt MA, Mamerow MM, Brown SA, Jolly CA. A Resilience Intervention in African American Adults With Type 2 Diabetes. The Diabetes Educator 2009;35(2):274-284. DOI: 10.1177/0145721708329698.
- 60. Davidson RJ, Kabat-Zinn J, Schumacher J, et al. Alterations in brain and immune function produced by mindfulness meditation. Psychosomatic medicine 2003;65(4):564-70. (In eng). DOI: 10.1097/01.psy.0000077505.67574.e3.
- 61. Larsen KL, Stanley EA. Mindfulness-based Mind Fitness Training (MMFT): Mindfulness training for highstress and trauma-sensitive contexts. Handbook of Mindfulness-Based Programmes: Routledge; 2019:53-63.
- 52. Jha AP, Zanesco AP, Denkova E, Rooks J, Morrison AB, Stanley EA. Comparing Mindfulness and Positivity Trainings in High-Demand Cohorts. Cognitive Therapy and Research 2020;44(2):311-326.
- 63. Lam SU, Kirvin-Quamme A, Goldberg SB. Overall and Differential Attrition in Mindfulness-Based Interventions: a Meta-Analysis. Mindfulness 2022. DOI: 10.1007/s12671-022-01970-z.
- 64. Stanic J, Barth J, Danon N, Bondolfi G, Jermann F, Eicher M. Adherence to standardized 8-week mindfulness-based interventions among women with breast or gynecological cancer: a scoping review. Journal of Psychosocial Oncology Research and Practice 2021;3(2) (<a href="https://journals.lww.com/jporp/Fulltext/2021/06000/Adherence\_to\_standardized\_8\_week\_mindfulness\_based.3.aspx">https://journals.lww.com/jporp/Fulltext/2021/06000/Adherence\_to\_standardized\_8\_week\_mindfulness\_based.3.aspx</a>).
- 65. Bachmann P, Finke JB, Rebeck D, et al. Test-retest reproducibility of a combined physical and cognitive stressor. Biological psychology 2019;148:107729. DOI: https://doi.org/10.1016/j.biopsycho.2019.107729.
- 66. O'Cathain A, Hoddinott P, Lewin S, et al. Maximising the impact of qualitative research in feasibility studies for randomised controlled trials: guidance for researchers. Pilot and Feasibility Studies 2015;1(1):32. DOI: 10.1186/s40814-015-0026-y.
- 67. Hsieh H-F, Shannon SE. Three Approaches to Qualitative Content Analysis. Qualitative Health Research 2005;15(9):1277-1288. DOI: 10.1177/1049732305276687.
- 68. Corp. I. IBM SPSS Statistics for Windows. 28 ed. Armonk, NY: IBM Corp; 2021.

Protocol version 2.4

- 69. Dhakal K. NVivo. Journal of the Medical Library Association 2022;110(2):270–272-270–272.
- 70. Atchley R, Ellingson R, Klee D, Memmott T, Oken B. A cognitive stressor for event-related potential studies: the Portland arithmetic stress task. Stress (Amsterdam, Netherlands) 2017;20(3):277-284. (In eng). DOI: 10.1080/10253890.2017.1335300.
- 71. Trottier JL, Oken BS. Mindfulness Meditation as a Stress Reactivity Intervention: An Event-Related Potential Study. 2017.

- 72. Johnstone JM, Roake C, Sheikh I, Mole A, Nigg JT, Oken B. School-based mindfulness intervention for stress reduction in adolescents: Design and methodology of an open-label, parallel group, randomized controlled trial. Contemporary clinical trials communications 2016;4:99-104.
- 73. Deyo RA, Diehr P, Patrick DL. Reproducibility and responsiveness of health status measures. Statistics and strategies for evaluation. Control Clin Trials 1991;12(4 Suppl):142s-158s. (In eng). DOI: 10.1016/s0197-2456(05)80019-4.
- 74. Fayers PM, Machin D. Quality of life: The assessment, analysis and reporting of patient-reported outcomes: John Wiley & Sons, 2015.
- 75. Eldridge SM, Chan CL, Campbell MJ, et al. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ (Clinical research ed) 2016;355:i5239. DOI: 10.1136/bmj.i5239.
- 76. Löwe B, Kroenke K, Herzog W, Gräfe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord 2004;81(1):61-6. (In eng). DOI: 10.1016/s0165-0327(03)00198-8.
- 77. Rush AJ, Trivedi MH, Carmody TJ, et al. Self-Reported Depressive Symptom Measures: Sensitivity to Detecting Change in a Randomized, Controlled Trial of Chronically Depressed, Nonpsychotic Outpatients. United Kingdom: Nature Publishing Group; 2005:405-416.
- 78. Hays RD, Anderson R, Revicki D. Psychometric considerations in evaluating health-related quality of life measures. Qual Life Res 1993;2(6):441-9. (In eng). DOI: 10.1007/bf00422218.
- 79. Middel B, van Sonderen E. Statistical significant change versus relevant or important change in (quasi) experimental design: some conceptual and methodological problems in estimating magnitude of intervention-related change in health services research. Int J Integr Care 2002;2:e15. (In eng). DOI: 10.5334/ijic.65.
- 80. Sivan M. Interpreting effect size to estimate responsiveness of outcome measures. Stroke 2009;40(12):e709; author reply e710-1. (In eng). DOI: 10.1161/strokeaha.109.566836.
- 81. Fok CC, Henry D. Increasing the Sensitivity of Measures to Change. Prev Sci 2015;16(7):978-86. (In eng). DOI: 10.1007/s11121-015-0545-z.
- 82. Lee AC, Driban JB, Price LL, Harvey WF, Rodday AM, Wang C. Responsiveness and Minimally Important Differences for 4 Patient-Reported Outcomes Measurement Information System Short Forms: Physical Function, Pain Interference, Depression, and Anxiety in Knee Osteoarthritis. J Pain 2017;18(9):1096-1110. (In eng). DOI: 10.1016/j.jpain.2017.05.001.
- 83. Revicki D, Hays RD, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. Journal of clinical epidemiology 2008;61(2):102-9. (In eng). DOI: 10.1016/j.jclinepi.2007.03.012.
- 84. Gallegos AM, Heffner KL, Cerulli C, Luck P, McGuinness S, Pigeon WR. Effects of mindfulness training on posttraumatic stress symptoms from a community-based pilot clinical trial among survivors of intimate partner violence. Psychological trauma: theory, research, practice and policy 2020;12(8):859-868. (In eng). DOI: 10.1037/tra0000975.